CLINICAL TRIAL: NCT03000855
Title: EUS - Guided Choledocho-duodenostomy Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Common Bile Duct Strictures. A Multi-centred Randomised Controlled Trial
Brief Title: EUS - Guided Choledocho-duodenostomy Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Common Bile Duct Strictures
Acronym: DRAMBO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tokyo Medical University (Other); Kinki University (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Honorary Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2016.193-T
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Malignant Biliary Obstruction
Keywords: Malignant biliary obstruction; EUS - guided choledocho-duodenostomy; ERCP with covered metallic stents
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECDS (Active Comparator): EUS-guided choledocho-duodenostomy
  Interventions: Procedure: EUS-guided choledocho-duodenostomy
- ERCP with CSEMS (Active Comparator): Endoscopic retrograde cholangiopancreatography with covered metallic stent
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography with covered metallic stent

INTERVENTIONS:
Procedure: EUS-guided choledocho-duodenostomy — The CBD would be identified by a linear echoendoscope and a suitable puncture site in the bulb of the duodenum would be located. The common bile duct would be punctured with a 19-gauge needle and the position would be confirmed by aspiration of bile and contrast injection. A 0.025" or 0.035" guide wire would be passed through the needle in to the CBD. A fully covered metal stent would then be inserted after track dilation.
  Arms: ECDS
Procedure: Endoscopic retrograde cholangiopancreatography with covered metallic stent — After cannulation of the CBD, a cholangiography would be performed to assess the diameter of the CBD, the length and position of the biliary stricture. The endoscopist would decide on the appropriate size of SEMS to be placed. The stents should be visible from the duodenal lumen after deployment.
  Arms: ERCP with CSEMS

SUMMARY:
EUS - guided choledocho-duodenostomy (ECDS) is an established option for bile duct drainage in unresectable malignant distal CBD strictures when endoscopic retrograde cholangiopancreatography (ERCP) fails. However, how primary ECDS compares with ERCP with covered self-expanding metallic stents (CSEMS) in unresectable malignant distal CBD strictures is uncertain.

The aim of the current study is to compare primary ECDS versus ERCP with CSEMS in unresectable malignant distal CBD strictures. We hypothesis that ECDS is associated with a higher 1-year stent patency rate.

DETAILED DESCRIPTION:
Malignant biliary obstruction is a common sequela of pancreatic cancers or distal bile duct cancers, and its development can hinder the use of chemotherapy, decrease patient quality of life and decrease survival. Malignant biliary obstruction is traditionally palliated with ERCP with metallic stent insertion. However, these stents are prone to obstruction due to tumour ingrowth. In addition, ERCP may not always be possible due to tumour obstruction and percutaneous biliary drainage may be required.

Recently, ECDS has been described as an alternative to percutaneous biliary drainage in patients with failed ERCP. The procedure is also associated with potential advantages as compared to conventional ERCP. In particular, the risk of tumour ingrowth into the stent placed after ECDS is low and stent patency rates may be better than ERCP. Thus, the aim of the current study is to compare primary ECDS versus ERCP with CSEMS in unresectable malignant distal CBD strictures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old with informed consent
* Histologically (preferred) or radiologically confirmed distal malignant bile duct tumors
* Inoperability by staging, comorbidities or patient wishes
* Distal tumors 2cm away from the portal hilum
* Bilirubin > 50umol/L at diagnosis

Exclusion Criteria:

* Multiple hepatic metastases with significant blockage of one or more liver segments (if no segment blockage, metastasis is not an exclusion criteria)
* Presence of main portal vein thrombosis
* Prior SEMS placement
* Intraductal papillary mucinous carcinomas
* Prior Billroth II or roux-en Y reconstruction
* History of bleeding disorder or use of anticoagulation
* Child's B/C cirrhosis
* Pregnancy
* Performance status ECOG ≥3 (confined to bed / chair > 50% waking hours)
* Presence of other malignancy
* Life expectancy < 3months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
stent patency rate | 1-year
  Stent dysfunction is defined as radiology or endoscopy confirmed stent obstruction.

SECONDARY OUTCOMES:
Technical success | 1year
  Technical success is defined as the ability to access and drain the CBD by placement of a stent.
Clinical success | 1 year
  Clinical success is defined as >30% drop in bilirubin levels
Adverse events | 30 days
  Adverse events related to the endoscopic procedures would be graded according to the lexicon of endoscopic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Teoh, FRCSEd(Gen, Principal Investigator — anthoyteoh@surgery.cuhk.edu.hk
Locations (6):
- Royal Prince Alfred Hospital, Sydney, Australia
- The University of Leuven, Leuven, Belgium
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China
- Aarhus University Hospital, Aarhus, Denmark
- Japan (2):
  - Tokyo Medical University Hospital, Tokyo
  - Wakayama Medical University School of Medicine, Wakayama

REFERENCES:
- [Derived] Teoh AYB, Napoleon B, Kunda R, Arcidiacono PG, Kongkam P, Larghi A, Van der Merwe S, Jacques J, Legros R, Thawee RE, Saxena P, Aerts M, Archibugi L, Chan SM, Fumex F, Kaffes AJ, Ma MTW, Messaoudi N, Rizzatti G, Ng KKC, Ng EKW, Chiu PWY. EUS-Guided Choledocho-duodenostomy Using Lumen Apposing Stent Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Trial (DRA-MBO Trial). Gastroenterology. 2023 Aug;165(2):473-482.e2. doi: 10.1053/j.gastro.2023.04.016. Epub 2023 Apr 28. PMID 37121331